CLINICAL TRIAL: NCT06149403
Title: A Multi-center, Randomized, Active Controlled Clinical Trial to Evaluate the Efficacy and Safety of OTL-203 in Subjects With Mucopolysaccharidosis Type I, Hurler Syndrome (MPS-IH) Compared to Standard of Care With Allogeneic Hematopoietic Stem Cell Transplantation (Allo-HSCT)
Brief Title: A Study to Investigate the Efficacy and Safety of OTL-203 in Subjects With MPS-IH Compared With Standard of Care With Allogeneic HSCT
Acronym: HURCULES
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Orchard Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OTL-203-02
Record Dates: First submitted 2023-11-17; First posted 2023-11-29 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: MPS-IH (Hurler Syndrome)
Keywords: MPS-IH; Hurler; MPS-I; Mucopolysaccharidoses; Mucopolysaccharidosis type I; Hurler syndrome; Mucopolysaccharidosis IH; Gene Therapy; Transplantation; Autologous Lentiviral vector
MeSH Terms: conditions — Mucopolysaccharidosis I; Mucopolysaccharidoses

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OTL-203 (Experimental): Eligible subjects randomized to Arm 1 will receive an intravenous (IV) infusion of OTL-203 gene therapy. Subjects will receive conditioning regimen with busulfan and fludarabine prior to OTL-203 infusion.
  Interventions: Genetic: Experimental: OTL-203
- Allo-HSCT (Active Comparator): Eligible subjects randomized to Arm 2 will receive allogeneic hematopoietic stem cell transplantation. Subjects will receive conditioning regimen with busulfan and fludarabine prior to allo-HSCT.
  Interventions: Genetic: Active Comparator: Allo-HSCT

INTERVENTIONS:
Genetic: Experimental: OTL-203 — Experimental: OTL-203: Autologous CD34+ enriched cell fraction that contains hematopoietic stem and progenitor cells transduced ex vivo using lentiviral vector encoding the human IDUA gene
  Arms: OTL-203
Genetic: Active Comparator: Allo-HSCT — Active Comparator: Allogeneic hematopoietic stem cell transplantation
  Arms: Allo-HSCT

SUMMARY:
A multi-center randomized clinical trial to compare OTL-203 (gene therapy) with stem cell transplant (standard of care) in patients with MPS-IH (Hurler syndrome).

DETAILED DESCRIPTION:
The study is a multi-center, randomized, active controlled clinical trial designed to evaluate the efficacy and safety of OTL-203 in patients with mucopolysaccharidosis type I, Hurler syndrome (MPS-IH) compared to standard of care with allogeneic hematopoietic stem cell transplantation (allo-HSCT). A total of 40 patients with a confirmed diagnosis of MPS-IH who meet the study inclusion criteria will be randomized to receive either OTL-203 or allo-HSCT. The trial will comprise of a screening, baseline, and treatment period, with a follow-up period of 5 years post-treatment, and primary analysis performed at 2 years follow-up of the last treated subject.

ELIGIBILITY:
Inclusion Criteria:

1. Norm-referenced cognitive standard score of ≥70 measured by age-appropriate cognitive domains of either Bayley Scale of Infant Development (BSID)-III or Wechsler Preschool and Primary Scale of Intelligence (WPPSI)-IV.
2. Confirmed laboratory diagnosis of MPS-IH as demonstrated by biallelic mutation(s) in the gene coding for IDUA enzyme
3. Final confirmation of MPS-IH diagnosis by a Diagnostic Review Committee (DRC).

Exclusion Criteria:

1. Previous allo-HSCT or gene therapy
2. Current enrollment or past treatment in any other interventional study/trial using a novel investigational agent and/or treated with prohibited medications listed in the protocol
3. Positivity to serological testing for Human Immunodeficiency Virus (HIV)-1 or HIV-2, Human T Lymphotropic Virus (HTLV)-1 or HTLV-2, Hepatitis B Virus (HBV) core, Hepatitis C Virus (HCV), mycoplasma, active tuberculosis (TB) and not meeting the microbiology biological screening requirements.
4. Malignant neoplasia (except local skin cancer).
5. Myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
6. History of uncontrolled seizures
7. Subjects with an active infection not responsive to treatment, end-organ damage, or any other disease that contraindicates performance of any of the procedures detailed in the protocol, or medical conditions or extenuating circumstances that, in the opinion of the Investigator, might compromise the subject's well-being or safety, or the interpretability of the subject's clinical data.
8. Subjects, who in the opinion of the Investigator, may not be able to comply with protocol requirements or cooperate fully with the study procedures and necessary long-term follow up

Ages: 28 Days to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 2 years
  Defined by events of death, rescue transplant, treatment failure, immunological complications, severe cognitive and/or growth impairment.

SECONDARY OUTCOMES:
Change from baseline to Year 2 in α-L-iduronidase (IDUA) activity in leukocytes | Day 30 and multiple visits up to 5 years post-treatment
  IDUA activity in leukocytes will be used to measure post-treatment systemic correction of the biochemical defect that causes the disease
Change from baseline to Year 2 in the ratio to the upper limit of normal (ULN) of urinary heparan sulfate levels | Day 30 and multiple visits up to 5 years post-treatment
  Urinary heparan sulfate levels will be used to measure post-treatment clearance of glycosaminoglycans accumulated within tissues and organs due to IDUA enzymatic deficiency
Safety of OTL-203 compared to allo-HSCT procedure | Up to 5 years post-treatment
  Measured by Overall incidence of adverse events (AEs) whether or not considered related to the study treatment, including conditioning regimen-related AEs, Study Procedure-related AEs, Disease-related AEs, Treatment related AEs, Serious adverse events (SAEs)
Malignancy or abnormal clonal proliferation (ACP) using different tests and procedures (e.g., general clinical evaluation, blood counts, and specialized assessments such as integration site analysis). | Up to 5 years post-treatment
  Malignancy or ACP due to insertional oncogenesis will be evaluated in subjects treated with OTL-203.
Replication Competent Lentivirus (RCL) | Up to 5 years post-treatment
  Presence of RCL will be evaluated in subjects treated with OTL-203
Immune response against IDUA enzyme | Up to 5 years post-treatment
  Anti-IDUA antibodies analysis will be evaluated in all subjects.

CONTACTS AND LOCATIONS:
Locations (5):
- University of Minnesota, Pediatrics, Minneapolis, Minnesota, United States
- Ospedale San Raffaele, Milan, Italy
- Netherlands (2):
  - Princess Maxima Center, Utrecht
  - UMC Utrecht, Utrecht
- Manchester University NHS Foundation Trust Blood and Marrow Transplant Programme, Royal Manchester Children's Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No